CLINICAL TRIAL: NCT03442322
Title: Optimizing Care for Patients With Dementia: A Comparison of Two Non-pharmacological Treatment Approaches
Brief Title: Optimizing Care for Patients With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Natalie Leland, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY19090117
Record Dates: First submitted 2018-01-31; First posted 2018-02-22 (Actual); Results first posted 2024-08-19 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer Disease
Keywords: long term care residents; nursing home care
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: This cluster pragmatic trial randomized eligible nursing homes to one of the two intervention arms according to the predetermined protocol to evaluate the effect of the facility-level intervention on resident (i.e. long term care residents living with Alzheimer's Disease or Related Dementia) and staff outcomes.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the treatment arm the facility is randomly assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transdisciplinary approach (Active Comparator): The transdisciplinary approach that is integrated across disciplines and provides core training for all providers, staff members, and stakeholders, using a common language to address care concerns and support continuity and sustainability
  Interventions: Other: transdisciplinary approach
- multidisciplinary approach (Active Comparator): The multidisciplinary approach that is problem-based and draws on the expertise of individual healthcare providers (e.g., occupational therapy) to address care concerns.
  Interventions: Other: multidisciplinary approach

INTERVENTIONS:
Other: transdisciplinary approach — This approach is integrated across disciplines and provides core training for all providers, staff members, and stakeholders, using a common language to address care concerns and support continuity and sustainability;
  Arms: transdisciplinary approach
Other: multidisciplinary approach — This is a problem-based approach that draws on the expertise of individual healthcare providers (e.g., occupational therapy) to address care concerns.
  Arms: multidisciplinary approach

SUMMARY:
Of the 1.4 million nursing home (NH) residents in long term care facilities, more than half have Alzheimer's disease or dementia. Due to changes in their familiar daily routines, difficulty expressing their thoughts or asking for what they need, and overstimulation (such as noise) or under stimulation (such as lack of activity), individuals with dementia often display disruptive behaviors like resisting help or continually repeating the same phrases. Medications are often prescribed to reduce agitation and aggressive behavior; however, these medications may not be effective and can have a negative impact on the individual. Therefore, families and other stakeholders strongly advocate the use of other types of approaches that focus on minimizing the cause of the behavior. Two facility-based methodologies include the transdisciplinary approach for integrated dementia care, which combines the expertise of all NH staff, who work together to build a common language and approach for each resident, and the multidisciplinary approach for problem-based dementia care, in which each staff member conducts individual assessments and makes discipline-specific recommendations. While prior research suggests that both of these facility-based approaches are useful, the circumstances under which each approach is most effective are not clear. This project will prospectively randomize 80 nursing homes to one of the two treatment arms to compare the effect of the transdisciplinary approach versus the multidisciplinary approach.

This study will examine the difference between the two comparators with respect to facility rates of medications dispensed to residents with dementia, leading to enhanced quality of life for the resident.

This project is important because it will address a key clinical dilemma NH staff face as they strive to optimize the use of alternative approaches to reduce disruptive behaviors in residents with dementia. Transforming the quality of dementia care in NHs and enhancing the quality of life of residents with dementia are high priorities for families and other advocates.

ELIGIBILITY:
Inclusion Criteria:

Eligible nursing home facilities will

* lack any existing dementia program targeting reduction of off-label psychotropic medication use
* each serve >60 long-term care residents with Alzheimer's or dementia
* meet Center for Medicare & Medicaid Services' minimum requirements for NHs (e.g., meeting the mandated number of hours of staff training on dementia care, performing regularly scheduled resident assessments).

Exclusion Criteria:

Facilities will be excluded if they have

* less than 60 long-stay residents
* an existing formal dementia care program in place
* an off-label psychotropic medication reduction program
* is located in a state that requires more than the Center for Medicare & Medicaid Services' minimum for staff training requirements on the topic of dementia care

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2022-07-26 (Actual); Study Completion 2022-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie E Leland, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Piersol CV, Martinez J, Chew F, Perry B, Leland NE. Understanding the Experiences of Family Caregivers of Nursing Home Residents With Dementia: A Grounded Theory Study. Gerontologist. 2024 Apr 1;64(4):gnad102. doi: 10.1093/geront/gnad102. PMID 37501632

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This mixed methods study used quantitative methods to examine nursing home resident outcomes of the two non-pharmacological approaches to dementia care (i.e., the primary study outcomes). Qualitative methods included one-time interviews with family caregivers and nursing home staff intended to understand their experiences with the two non-pharmacological approaches. Flow chart below reflects the participating nursing homes (i.e., units) and their residents with dementia (i.e. participants).
Units Other Than Participants: Nursing homes
Period: Overall Study
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Started | 1291; 17 Nursing homes | 3206; 36 Nursing homes
6-month Outcome | 793; 17 Nursing homes | 1905; 36 Nursing homes
12-month Outcome | 658; 16 Nursing homes | 1693; 36 Nursing homes
Completed (This is the 18-month outcome) | 526; 16 Nursing homes | 1420; 36 Nursing homes
Not Completed | 765; 1 Nursing homes | 1786; 0 Nursing homes

BASELINE CHARACTERISTICS:
Population: This was a nursing home-level analysis, therefore not all participants were in the sample during the baseline period. Participants (i.e., nursing home residents) were included if they met the study criteria based on age, dementia status, and long-term nursing home residence, but could be included in the sample at any point of the study. Thus, there were participants who were in the study sample (and reflected in the flow overview), but were not in the study sample during the baseline period.
Units Other Than Participants: Nursing homes
Groups:
- Transdisciplinary Approach: This approach is integrated across disciplines and provides core training for all providers, staff members, and stakeholders, using a common language to address care concerns and support continuity and sustainability.
- Total: Total of all reporting groups
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach | Total
Number analyzed (Participants) | 759 | 1969 | 2728
Number analyzed (Nursing homes) | 17 | 36 | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 84.2 (8.1) | 84.9 (8.4) | 84.7 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 532 | 1469 | 2001
  Male | 227 | 500 | 727
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 622 | 1589 | 2211
  Black, non-Hispanic | 45 | 244 | 289
  Hispanic | 69 | 91 | 160
  Asian | 9 | 6 | 15
  Other | 14 | 39 | 53
Cognitive Function Scale [Count of Participants; unit: Participants]
  Cognitively Intact | 80 | 219 | 299
  Mildly impaired | 123 | 369 | 492
  Moderately impaired | 427 | 1138 | 1565
  Severely impaired | 129 | 243 | 372
Number of Nursing Home Beds [Mean (Standard Deviation); unit: certified beds] | 118.6 (50.2) | 119.9 (38.0) | 119.5 (41.8)
Nursing Home Occupancy Rate [Mean (Standard Deviation); unit: # of occupied beds/ # of certified beds] | 0.87 (0.1) | 0.87 (0.1) | 0.87 (0.1)
CMS Nursing Home Rating [Mean (Standard Deviation); unit: units on a scale] — This is the Centers for Medicare and Medicaid (CMS) 5-Star Rating for nursing homes, which is a composite measure of quality reflecting state survey performance, staffing, and quality. The measure ranges from 1 to 5, with a score of 1 indicating low care quality and 5 indicates high care quality.
  units on a scale
    State Survey | 2.6 (1.2) | 2.7 (1.2) | 2.7 (1.2)
    Staffing Levels | 3.1 (0.7) | 2.7 (1.0) | 2.8 (0.9)
    Quality of Care | 3.5 (1.1) | 3.6 (1.1) | 3.5 (1.1)
Quality Measures [Mean (Standard Deviation); unit: percentage of long-stay residents]
  increased in need for help with ADL | 18.3 (6.7) | 17.3 (5.4) | 17.6 (5.8)
  had pressure ulcer | 8.8 (3.7) | 8.3 (3.7) | 8.5 (3.7)
  lost too much weight | 5.6 (2.5) | 7.3 (3.5) | 6.8 (3.3)
  had catheter inserted and left in bladder | 1.4 (1.2) | 1.3 (1.4) | 1.3 (1.3)
  had urinary tract infection | 2.9 (2.5) | 2.1 (1.6) | 2.4 (1.9)
  have depressive symptoms | 4.6 (5.7) | 3.6 (4.1) | 3.8 (4.6)
  were physically restrained | 0.1 (0.3) | 0.2 (0.5) | 0.1 (0.4)
  had fall(s) with injury | 4.2 (1.9) | 3.1 (2.5) | 3.5 (2.4)
  received antipsychotic medication | 12.7 (3.9) | 13.4 (6.4) | 13.2 (5.7)
  ability to move independently worsened | 21.2 (9.9) | 21.3 (7.8) | 21.2 (8.4)
  received antianxiety/hypnotic medication | 22.4 (7.3) | 21.4 (11.5) | 21.7 (10.3)

OUTCOME MEASURES:

1. Primary Outcome: Dispensing of Psychotropic Medications
Description: Percentage of nursing home residents with dementia who received one or more antipsychotic medication over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: Population includes all nursing home residents with dementia in participating nursing homes with valid data in the Minimum Data Set (MDS) assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 742 | 1787
Participants | 161 | 315
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — Given that we found baseline differences in resident characteristics and outcomes, we implemented a difference-in-differences model for all outcomes; p = 0.492, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = 1.25

2. Primary Outcome: Dispensing of Psychotropic Medications
Description: Percentage of nursing home residents with dementia who received one or more antipsychotic medication over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: Population includes all nursing home residents with dementia in participating nursing homes (NHs) with valid data in the Minimum Data Set (MDS) assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 606 | 1564
Participants | 125 | 289
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.765, Regression, Linear; All regressions controlled for resident characteristics, nursing home staffing, resident COVID cases, and nursing home fixed effects; Difference-in-Difference estimator = -0.73

3. Primary Outcome: Dispensing of Psychotropic Medications
Description: Percentage of nursing home residents with dementia who received one or more antipsychotic medication over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: Population includes all nursing home residents with dementia in participating NHs with valid data in the Minimum Data Set (MDS) assessments.
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 487 | 1303
Participants | 107 | 227
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.808, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 0.77

4. Primary Outcome: Behavioral Symptoms
Description: Percentage of nursing home residents with dementia who had behavioral symptoms over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 788 | 1889
Participants | 143 | 334
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.108, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = 3.86

5. Primary Outcome: Behavioral Symptoms
Description: Percentage of nursing home residents with dementia who had behavioral symptoms over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 648 | 1654
Participants | 104 | 299
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.411, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 2.59

6. Primary Outcome: Behavioral Symptoms
Description: Percentage of nursing home residents with dementia who had behavioral symptoms over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 521 | 1392
Participants | 68 | 232
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.981, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -0.08

7. Primary Outcome: Wandering
Description: Percentage of nursing home residents with dementia who had wandering over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 788 | 1889
Participants | 88 | 117
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.020, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = 3.51

8. Primary Outcome: Wandering
Description: Percentage of nursing home residents with dementia who had wandering over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 648 | 1653
Participants | 52 | 116
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.299, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 1.62

9. Primary Outcome: Wandering
Description: Percentage of nursing home residents with dementia who had wandering over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 521 | 1393
Participants | 38 | 98
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.389, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 1.68

10. Primary Outcome: Rejection of Care
Description: Percentage of nursing home residents with dementia who had rejection of care over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 788 | 1889
Participants | 131 | 302
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.389, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = -2.14

11. Primary Outcome: Rejection of Care
Description: Percentage of nursing home residents with dementia who had rejection of care over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 648 | 1653
Participants | 75 | 282
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.043, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -5.95

12. Primary Outcome: Rejection of Care
Description: Percentage of nursing home residents with dementia who had rejection of care over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 521 | 1393
Participants | 59 | 217
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.279, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -3.91

13. Secondary Outcome: Unintended Weight Loss
Description: Percentage of nursing home residents with dementia who had unintended weight loss over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 781 | 1884
Participants | 125 | 302
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.728, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = 0.92

14. Secondary Outcome: Unintended Weight Loss
Description: Percentage of nursing home residents with dementia who had unintended weight loss over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 640 | 1651
Participants | 132 | 395
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.490, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -1.75

15. Secondary Outcome: Unintended Weight Loss
Description: Percentage of nursing home residents with dementia who had unintended weight loss over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 517 | 1394
Participants | 137 | 294
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.232, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 4.44

16. Secondary Outcome: Falls
Description: Percent of nursing home residents with dementia who had falls over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 785 | 1887
Participants | 326 | 750
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.708, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = 1.11

17. Secondary Outcome: Falls
Description: Percent of nursing home residents with dementia who had falls over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 644 | 1652
Participants | 274 | 700
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.775, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 1.00

18. Secondary Outcome: Falls
Description: Percent of nursing home residents with dementia who had falls over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 520 | 1387
Participants | 246 | 614
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.584, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = 1.77

19. Secondary Outcome: Depressive Symptoms
Description: Percent of nursing home residents with dementia who had depressive symptoms over Months 1-6 of Intervention
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 680 | 1676
Participants | 37 | 90
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.898, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = -0.25

20. Secondary Outcome: Depressive Symptoms
Description: Percent of nursing home residents with dementia who had depressive symptoms over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 545 | 1408
Participants | 24 | 95
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.217, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -2.79

21. Secondary Outcome: Depressive Symptoms
Description: Percent of nursing home residents with dementia who had depressive symptoms over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 437 | 1195
Participants | 20 | 59
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.560, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -1.39

22. Secondary Outcome: Physical Restraints Use
Description: Percent of nursing home residents with dementia who had physical restraint use over Months 1-6 of Intervention.
Time Frame: 6-month period (months 1-6)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 786 | 1887
Participants | 3 | 102
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.277, Regression, Linear; All regressions controlled for resident characteristics and nursing home fixed effects; Difference-in-Difference estimator = -3.08

23. Secondary Outcome: Physical Restraints Use
Description: Percent of nursing home residents with dementia who had physical restraint use over Months 7-12 of Intervention.
Time Frame: 12-month period (months 7-12)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 644 | 1652
Participants | 4 | 91
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.400, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -2.53

24. Secondary Outcome: Physical Restraints Use
Description: Percent of nursing home residents with dementia who had physical restraint use over Months 13-18 of Intervention.
Time Frame: 18-month period (months 13-18)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
Number analyzed (Participants) | 520 | 1387
Participants | 0 | 70
Statistical Analysis 1: Comparison: Transdisciplinary Approach vs Multidisciplinary Approach; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.303, Regression, Linear; [statistical method as in outcome 2, analysis 1]; Difference-in-Difference estimator = -3.18

ADVERSE EVENTS:
Time Frame: This pragmatic clinical trial was embedded into the workflow of the nursing homes. Our intervention was about training staff about dementia knowledge. We were not intervening at patient level, thus adverse outcomes were not relevant.
Description: This pragmatic clinical trial was embedded into the workflow of the nursing homes. Our intervention was about training staff about dementia knowledge. We were not intervening at patient level, thus adverse outcomes were not relevant.
Arm/Group | Transdisciplinary Approach | Multidisciplinary Approach
All-Cause Mortality (participants affected / at risk) | 0/1291 | 0/3206
Serious Adverse Events (participants affected / at risk) | 0/1291 | 0/3206
Other Adverse Events (participants affected / at risk) | 0/1291 | 0/3206

LIMITATIONS AND CAVEATS:
We were only able to assess post-training outcomes for 6 months prior to COVID-19 and it is possible that nursing homes would have achieved different outcomes after this initial start-up period. Similarly, the comparative effectiveness of the care approaches in 12- and 18-month follow-up period were confounded by the effects of COVID-19. Finally, the use of antipsychotic medication outcome was collected with a 7-day look back period, which may have resulted in underreporting.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/22/NCT03442322/Prot_SAP_000.pdf